CLINICAL TRIAL: NCT03000140
Title: Health Status Factors Predicting Responses to Long-Term Training: Effects of 16-Week High-Intensity Interval Training on Pre-Hypertensive Subjects
Brief Title: High-Intensity Interval Training on Pre-Hypertensive Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Healthcare Center Tomas Rojas (Other); University of Los Ríos (Unknown); Universidad Pública de Navarra (Other); Universidad del Rosario (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Number 03052015
Record Dates: First submitted 2016-12-17; First posted 2016-12-21 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Metabolism Disorder; Hypertension
MeSH Terms: conditions — Metabolic Diseases; Hypertension | interventions — High-Intensity Interval Training; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Intensity Interval Training (Experimental): Cycling on cycle ergometers (OXFORDTM, model BE2601, OXOFORD Inc, Santiago, Chile) for 1 min at a subjective intensity of 8-10 points of the modified Borg scale of 1-10 points, and interspersed by inactive (without movement over the bicycle) of 2 minutes as recovery period.
  Interventions: Behavioral: High Intensity Interval Training
- Control group (Active Comparator): Pre-hypertensive group was compared with healthy groups in the 2 manin variables systolic/diastolic blood pressure, as well as in other co-variables in pre-post changes. Thus, after the training intervention, and following the R and NR classification, we will compare the NR prevalence between both Pre-hypertensive and Healthy group.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: High Intensity Interval Training — High Intensity Interval Training pre-hypertensive group; Exercise will be performed at three sessions per week. All sessions will be supervised by an exercise physiologist during 16 weeks.
  Arms: High Intensity Interval Training
Behavioral: Control group — Moderade Intensity Interval Training pre-hypertensive group; Exercise will be performed at three sessions per week. All sessions will be supervised by an exercise physiologist during 16 weeks.
  Arms: Control group

SUMMARY:
Despite exercise training decrease blood pressure in 'average' terms, there is a wide interindividual variability after exercise training, being yet unknown what mode of exercise (e.g. endurance, strength, concurrent, or high intensity interval training) produce more/less non-responder (NR) prevalence (i.e., percentage of subjects who experienced a non-change/worsened response after training in some outcome).

DETAILED DESCRIPTION:
Despite exercise training decrease blood pressure in 'average' terms, there is a wide interindividual variability after exercise training, being yet unknown what mode of exercise (e.g. endurance, strength, concurrent, or high intensity interval training) produce more/less non-responder (NR) prevalence (i.e., percentage of subjects who experienced a non-change/worsened response after training in some outcome).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Interested in improving health and fitness;
* Systolic blood pressure > 120 mmHg and < 140 mmHg, and/or DBP ≥ 80 and < 90 mmHg according with standard classification;
* No drug therapy during the previous 3 months;
* Body mass index (BMI) 25 and 35 kg/m2); (c) physically inactive (according to the International Physical Activity Questionnaire previously validated in Chilean population)
* Normal /mild altered lipid profile (total cholesterol [TC] ~200 and ≤250 mg/dL, low-density lipids [LDL-C] ~140 mg/dL and ≤200 mg/dL, high-density lipids [HDL-C] ≥20 and ~40 mg/dL, triglycerides ~150 and ≤250 mg/dL) according with standard classification.

Exclusion Criteria:

* Cardiovascular contraindications to exercise histories of stroke;
* Asthma and chronic obstructive pulmonary disease;
* Musculoskeletal disorder such as low back pain;
* Smokers in the last 3 months were not included in the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in systolic blood pressure and diastolic blood pressure | Baseline and 16 weeks immediately after the interventions ends
  After this, we calculated the delta changes in both variables and classified to all subjects in responders (R) and non-responders (NR) to decrease systolic or diastolic blood pressure.

SECONDARY OUTCOMES:
Change from Baseline in body mass | Baseline and 16 weeks immediately after the interventions ends
Change from Baseline in body mass index | Baseline and 16 weeks immediately after the interventions ends
  BMI will be calculated as the body weight in kilograms divided by the square of the height in meters.
Change from Baseline in waist circumference | Baseline and 16 weeks immediately after the interventions ends
Change from Baseline in fat mass | Baseline and 16 weeks immediately after the interventions ends
Change from Baseline in heart rate at rest | Baseline and 16 weeks immediately after the interventions ends
  Baseline and 16 weeks immediately after the interventions ends
Change from Baseline in fasting glucose | Baseline and 16 weeks immediately after the interventions ends
Change from Baseline in lipids | Baseline and 16 weeks immediately after the interventions ends
  Lipid profile (low-density cholesterol, total cholesterol, high-density cholesterol and triglycerides)
Change from Baseline in one maximum repetition strength test of leg-extension exercise | Baseline and 16 weeks immediately after the interventions ends

CONTACTS AND LOCATIONS:
Locations (1):
- Cristian Alvarez, Osorno, Chile

REFERENCES:
- [Derived] Alvarez C, Ramirez-Campillo R, Cristi-Montero C, Ramirez-Velez R, Izquierdo M. Prevalence of Non-responders for Blood Pressure and Cardiometabolic Risk Factors Among Prehypertensive Women After Long-Term High-Intensity Interval Training. Front Physiol. 2018 Oct 23;9:1443. doi: 10.3389/fphys.2018.01443. eCollection 2018. PMID 30405426